CLINICAL TRIAL: NCT04432571
Title: An Adaptive Strategy for Preventing and Treating Lapses of Retention in HIV Care for Adolescents
Brief Title: ADAPT for Adolescents Adolescents
Acronym: A4A
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Colorado, Denver (Other); University of California, San Francisco (Other); University of California, Berkeley (Other); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201910133
Record Dates: First submitted 2020-06-04; First posted 2020-06-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: HIV/AIDS
Keywords: Adolescents; Retention; Engagement in Care; Lost to follow-up; Kenya; Adaptive strategies; Sequentially randomized trial; Sequential Multiple Assignment Randomized Trial
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SOC-REC/SOC-OIC (Active Comparator): Standard of care - routine education and counseling (SOC-REC)/SOC-Outreach and Intensified Counseling (OIC)
  Interventions: Behavioral: SOC-REC/SOC-OIC
- SOC-REC/CCT (Experimental): SOC-REC/Conditional Cash Transfer (CCT)
  Interventions: Behavioral: SOC-REC/CCT
- SOC-REC/IP-NAV (Experimental): SOC-REC/In-Person Peer Navigation (IP-NAV)
  Interventions: Behavioral: SOC-REC/IP-NAV
- E-NAV/SOC-OIC (Experimental): Electronic Navigation/SOC-OIC
  Interventions: Behavioral: E-NAV/SOC-OIC
- E-NAV/CCT (Experimental): E-Nav/Conditional cash transfer
  Interventions: Behavioral: E-NAV/CCT
- E-NAV/IP-NAV (Experimental): E-Nav/In-Person Peer Navigation
  Interventions: Behavioral: E-Nav/IP-NAV

INTERVENTIONS:
Behavioral: SOC-REC/SOC-OIC — Standard of care - routine education and counseling (SOC-REC)/SOC-Outreach and Intensified Counseling (OIC). SOC-REC is a stage 1 intervention to prevent lapses in HIV engagement through routine care. If an adolescent (1) misses an appointment >14 days, or (2) who have unsuppressed HIV RNA as per current MOH viral load threshold or (3) clinically documented non-adherence after >3 months of treatment he/she is re-randomized to a stage 2 intervention. SOC-OIC is a stage 2 intervention to treat lapses in HIV engagement through routine care which may include tracing and counseling to return to the clinic.
  Other Names: Standard of care-routine education and counseling/Outreach and Intensified Counselling
  Arms: SOC-REC/SOC-OIC
Behavioral: SOC-REC/CCT — SOC-REC/Conditional Cash Transfer (CCT). SOC-REC is a stage 1 intervention to prevent lapses in HIV engagement through routine care. If an adolescent (1) misses an appointment >14 days, or (2) who have unsuppressed HIV RNA as per current MOH viral load threshold or (3) clinically documented non-adherence after >3 months of treatment he/she is re-randomized to a stage 2 intervention. CCT is a stage 2 intervention to treat lapses in HIV engagement by providing a small cash incentive for on-time clinic attendance and/or viral load suppression (following per current MOH guidelines).
  Other Names: Standard of care-routine education and counseling/Conditional Cash Transfer
  Arms: SOC-REC/CCT
Behavioral: SOC-REC/IP-NAV — SOC-REC/In-Person Peer Navigation (IP-NAV). SOC-REC is a stage 1 intervention (routine care) to prevent lapses in HIV engagement. If an adolescent (1) misses an appointment >14 days, or (2) who have unsuppressed HIV RNA as per current MOH viral load threshold or (3) clinically documented non-adherence after >3 months of treatment he/she is re-randomized to a stage 2 intervention. IP-NAV is a stage 2 intervention to treat lapses in HIV engagement. Trained peer navigators will develop rapport with the participants and provide psychosocial support, case management, and assess retention and adherence barriers in a systematic manner and work with the participant to develop social support and clear, feasible plans to address barriers. The peer navigator will meet with the participant at least monthly, and no more than weekly, until HIV care engagement is demonstrated.
  Other Names: Standard of care-routine education and counseling/In-Person Peer Navigation
  Arms: SOC-REC/IP-NAV
Behavioral: E-NAV/SOC-OIC — E-Nav is a stage 1 intervention to prevent lapses in HIV engagement. Trained e-peer navigators will develop rapport and provide support through phone calls and/or patient preferred social media platforms. They will meet once in person and then weekly electronically for 8 weeks, and then monthly. If an adolescent (1) misses an appointment >14 days, or (2) who have unsuppressed HIV RNA as per current MOH viral load threshold or (3) clinically documented non-adherence after >3 months of treatment he/she is re-randomized to a stage 2 intervention. SOC-OIC is a stage 2 intervention to treat lapses in HIV engagement through routine care which may include tracing and counseling to return to the clinic.
  Other Names: Electronic-Navigation/SOC-Outreach and Intensified Counseling
  Arms: E-NAV/SOC-OIC
Behavioral: E-NAV/CCT — E-Nav is a stage 1 intervention to prevent lapses in HIV engagement. Trained e-peer navigators will develop rapport and provide support through phone calls and/or patient preferred social media platforms. They will meet once in person and then weekly electronically for 8 weeks, and then monthly. If an adolescent (1) misses an appointment >14 days, or (2) who have unsuppressed HIV RNA as per current MOH viral load threshold or (3) clinically documented non-adherence after >3 months of treatment he/she is re-randomized to a stage 2 intervention. CCT is a stage 2 intervention to treat lapses in HIV engagement by providing a small cash incentive for on-time clinic attendance and/or viral load suppression (following current MOH guidelines).
  Other Names: Electronic-Navigation/Conditional cash transfer
  Arms: E-NAV/CCT
Behavioral: E-Nav/IP-NAV — E-Nav is a stage 1 intervention to prevent lapses in HIV engagement. Trained e-peer navigators will develop rapport and provide support through phone calls and/or patient preferred social media platforms. They will meet once in person and then weekly electronically for 8 weeks, and then monthly. If an adolescent (1) misses an appointment >14 days, or (2) has unsuppressed HIV RNA as per current MOH viral load threshold or (3) clinically documented non-adherence after >3 months of treatment he/she is re-randomized to a stage 2 intervention. IP-NAV is a stage 2 intervention to treat lapses in HIV engagement by providing in person navigation and counseling to a cash incentive for on-time clinic attendance and/or viral load suppression (MOH guidelines). Trained peer navigators will provide psychosocial support, case management, assess retention and adherence barriers in a systematic manner and work with the participant to develop social support and clear, feasible plans to address barriers
  Other Names: Electronic-Navigation/In-Person Peer Navigation
  Arms: E-NAV/IP-NAV

SUMMARY:
Adolescents and young adults (AYA) with HIV face unique challenges to engagement in care and their ability to achieve optimal health outcomes. The investigators hypothesize that developmentally-tailored behavioral interventions will improve engagement in HIV care and viral suppression (per current MOH guidelines) among AYA with HIV in Kenya. This two stage study will initially randomize 880 AYA with HIV to either standard of care (SOC) or electronic navigation to prevent treatment lapse. Participants who have a lapse will be re-randomized to SOC, in-person peer navigation, or conditional cash transfers. Formative work will be conducted initially to tailor the interventions to AYA and then later to assess AYA perception, experience, and satisfaction with the interventions. We will evaluate the most effective and cost-effective intervention and sequence of interventions to inform HIV program managers, public policy makers, and other key stakeholders the best approaches to improve engagement of care of AYA with HIV.

DETAILED DESCRIPTION:
While the global response to HIV has reached close to 20 million persons with life-saving antiretroviral therapy (ART) and saved upwards of 60 million life-years, progress has been uneven and adolescents and young adults (AYA) aged 14-24 years represent a key group left behind. Compared to adults, AYA with HIV face more numerous, more diverse and more intense barriers to adherence and retention. The investigators will utilize a SMART study design in two stages among 880 AYA with HIV in Kenya to improve retention and viral suppression per the current MOH guidelines. In stage 1 AYA will be randomized 1:1 to either (1) standard of care education or counseling vs. (2) electronic navigation. Participants who do well (no lapses in retention, medication pick up and viral suppression) will be maintained on these low-intensity interventions, whereas those who fail will be re-randomized a second time to one of three re-engagement interventions (stage 2): (1) standard of care tracing, (2) a conditional cash transfer and (3) in-person peer navigation. The primary outcomes include (1) for prevention: lapse in engagement or viral non-suppression following current MOH guidelines; (2) for re-engagement: viral suppression six months after re-randomization; and (3) across six strategies: sustained viral suppression and sustained engagement in care at two years. The investigators anticipate that enrolling 880 AYA will result in 99% power to detect a 15% difference in the primary outcome between intervention groups. The investigators believe this study will yield evidence specific to AYA with HIV, quantify the relative magnitude of different sequenced interventions, capture the costs, and have direct relevance for public health programming to end the AIDS epidemic through engaging adolescents and young adults with HIV.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection, on or initiating ART,
* 14-24 years of age,
* Living > 6 months in Kisumu County, Kenya in previous year,
* Capable of informed consent (> 18 years) or with a legal caregiver available for consent (14-<18 years),
* Access to a cell phone,
* Ability to read or be read short message service (SMS) messages,
* Willingness to be contacted by clinic upon missed appointment,
* For AYA who report phone sharing must have disclosed to the person sharing the phone.
* Additionally, we will include AYA who are aware of their HIV status or whose caregivers agree to assisted disclosure.

Exclusion Criteria:

* AYA who participated in ADAPT-R,
* Those planning to move out of Kisumu County, those acutely ill and requiring hospitalization,
* Those who report sharing phones but have not disclosed to the person sharing the phone

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 880 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2025-09-13 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Care engagement failure | 24 months
  Experiencing any of the following three events within the first year of follow-up: lapse in retention (defined as 14 days late for a scheduled visit) or unsuppressed HIV RNA following current MOH guidelines during routine monitoring, or death.
Re-engagement | 24 months
  Viral suppression (per current MOH guidelines) six months after re-randomization
Sustained viral suppression and engagement in care | 24 months
  Sustained viral suppression (per current MOH guidelines) and sustained engagement in care at 24 months

SECONDARY OUTCOMES:
Compare survival between arms | 24 months
  Use log rank test to compare survival curves between arms
Explore alternative outcome definitions: Mean visit adherence | 24 months
  mean number of scheduled clinic visits attended
Explore alternative outcome definitions: Medication possession ratio | 24 months
  Proportion of scheduled pharmacy/medication visits attended
Explore alternative outcome definitions: HIV RNA levels | 24 months
  Viral suppression threshold (following current MOH guidelines)
Composite of time to return and time to viral resuppression | 24 months
  Composite of time to return for the subset of patients failing Stage 1 treatments through missed visits, and time to viral resuppression for those who failed through an elevated viral load
Cost effectiveness | 24 months
  We will compute unit cost for intervention activity and use information on activities for each participant to compute intervention cost per participant for each intervention strategy.
Qualitative evaluation of how interventions work | 24 months
  Qualitative methods will be used to identify major themes to understand how interventions worked (or did not work).

CONTACTS AND LOCATIONS:
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya

REFERENCES:
- [Derived] Abuogi LL, Kulzer JL, Akama E, Odeny TA, Eshun-Wilson I, Petersen M, Shade SB, Montoya LM, Beres LK, Iguna S, Adhiambo HF, Osoro J, Opondo I, Sang N, Kwena Z, Bukusi EA, Geng EH. Adapt for Adolescents: Protocol for a sequential multiple assignment randomized trial to improve retention and viral suppression among adolescents and young adults living with HIV in Kenya. Contemp Clin Trials. 2023 Apr;127:107123. doi: 10.1016/j.cct.2023.107123. Epub 2023 Feb 20. PMID 36813086